CLINICAL TRIAL: NCT03379636
Title: Immediate and Short-term Effects of Kinesiotaping on Muscular Activity, Mobility, Strength and Pain After Rotator Cuff Surgery: A Cross-over Clinical Trial
Brief Title: Effects of Kinesiotaping on Muscular Activity, Mobility, Strength and Pain After Rotator Cuff Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CliniqueRR-006
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Rotator Cuff Tear
Keywords: Athletic tape; Electromyography; Rehabilitation; Shoulder
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: All subjects were tested without tape, with kinesiotape (KT) and with a sham tape (ST). KT and ST were applied in a randomized order.
  The sequence always began with the NT condition. Then the two tapes were applied in a randomized order and the subjects repeated the same procedure. Group allocation, KT vs ST group, corresponded to the last tape the subject received and had to wear for the next three days. A computer block (n=8) randomization process was performed and sealed opaque envelopes were used.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The physiotherapist who applied the tape was not blinded but he did not participate in outcome assessment. The main investigator who collected the data was blind as subjects wore a long-sleeve shirt which hid the tape and the tape was administered behind a folding screen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no tape (No Intervention): tests are realised without any shoulder tape
- kinesiotape (Experimental): tests are realised with a kinesiotape applied according to Dr Kase model, over the deltoid muscle and over the acromioclavicular joint
  Interventions: Device: kinesiotape
- sham tape (Sham Comparator): tests are realised with a sham tape, applied transversally under the deltoid tuberosity with no tension and with no direct influence on shoulder area
  Interventions: Device: sham tape

INTERVENTIONS:
Device: kinesiotape — Application of an elastic beige 5-cm width Leukotape®K (BSN medical, Germany). The first strip, a Y-strip, was applied with 10% to 15% of tension over the deltoid muscle, from origin to insertion with the first tail along the anterior deltoid while the arm was externally rotated and horizontally abducted. The second tail was applied along the posterior deltoid with the arm horizontally adducted and internally rotated. A second strip, an I-strip, was applied for mechanical correction, transversally in the sagittal plane over the acromioclavicular joint with a downward pressure applied to the KT, the arm being at trunk side
  Arms: kinesiotape
Device: sham tape — a rigid Leukotape®Classic (BSN medical, Germany) was used. A 5-cm strip was applied transversally under the deltoid tuberosity with no tension and with no direct influence on shoulder area.
  Arms: sham tape

SUMMARY:
Kinesiotape (KT) is widely used in musculoskeletal rehabilitation as an adjuvant to treatment but minimal evidence supports its use. The aim of this study is to determine the immediate and short-term effects of shoulder KT on muscular activity, mobility, strength and pain after rotator cuff surgery. Our hypotheses were that KT should not improve muscle function, mobility, strength or pain in a clinically meaningful way.

Methods: Thirty-nine subjects with shoulder rotator cuff surgery were tested 6 and 12 weeks post-surgery, without tape, with KT and with a sham tape (ST). KT and ST were applied in a randomized order. For each condition, muscular activity of upper trapezius, three parts of deltoid and infraspinatus during shoulder flexion, range of motion (ROM) and pain intensity were assessed. At 12 weeks, isometric strength at 90° of shoulder flexion, with related muscular activity and pain intensity were also measured. Subjects maintained the last tape applied for three days and recorded pain intensity at wake-up and during the day.

DETAILED DESCRIPTION:
Sample size was calculated a priori using STATA Version 13.1 software (StataCorp, College Station, USA). Based on data of muscular activity from the article of Hsu et al 20 and considering a statistical power of 80% and a Type I error of .05, a need for at least 36 subjects was necessary to highlight a group difference. We finally enrolled 39 subjects between January 2013 and October 2016. Informed written consent was obtained from all subjects and all rights of the participants were protected.

Testing procedure:

Subjects were invited to come at the Clinique romande de réadaptation in Sion (Switzerland) on two occasions: 6 and 12 weeks after their surgery. Each time, they first filled the French version of the quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire in order to assess their physical function and symptoms. This 11-item questionnaire is valid, reliable and responsive in shoulder disorders.14, 17 They also estimated their pain intensity at rest using a 100-mm visual analogue scale (VAS).

A baseline measurement was then realized, without any tape (NT). The subjects were seated on a chair without resting on the backrest, the arms along the body. Shoulder rotation was neutral, elbow extended and forearm in neutral position. The subjects had to lift their arm in the sagittal plane as high as possible, hold the position for 5 seconds and then return at initial position. The movement was repeated once after one minute rest.

During the second session, at 12 weeks, the subjects realized in addition a maximal voluntary isometric contraction measure (MVIC). The measure was realized at 90° of shoulder flexion, neutral rotation, elbow extended, pronation of the forearm and fist closed. The strap of the dynamometer was applied at the level of the wrist.5 The subjects had to develop the maximal force during a 5-seconds period. After one minute rest, a second trial took place. The whole session was videotaped for further analysis. At the end of the testing sessions, the subjects were instructed not to remove the last tape applied for 72 hours.

The sequence always began with the NT condition. Then the two tapes were applied in a randomized order and the subjects repeated the same procedure. Group allocation, KT vs ST group, corresponded to the last tape the subject received and had to wear for the next three days. A computer block (n=8) randomization process was performed and sealed opaque envelopes were used. The physiotherapist who applied the tape was not blinded but he did not participate in outcome assessment. The main investigator (first author) who collected the data was blind as subjects wore a long-sleeve shirt which hid the tape and the tape was administered behind a folding screen.

Statistical analysis:

Comparisons between baseline characteristics of the two groups were computed using nonparametric tests comparing the medians for continuous variables or chi-squared tests for categorical variables.

The outcome variables measured during the mobility and the strength tests were compared between the three taping conditions. For the VAS outcomes during the three days after tape application, comparisons were realized between KT and ST solely. As the distributions of the outcome variables were not normal, nonparametric tests comparing the medians were performed. All analyses were done using Stata 13.1 software.

As multiple comparisons were realized, the level of statistical significance was set at P<.017 (.05/3) for the comparisons between the three conditions of tape (comparison of NT vs KT, NT vs ST, KT vs ST). For comparison between KT group and ST group only, the level of significance was set at P<.05.

ELIGIBILITY:
Inclusion Criteria:

* adult subject who had a surgery less than 6 weeks ago after a shoulder rotator cuff tear

Exclusion Criteria:

* re-tear of the rotator cuff, associated neurological lesion, concomitant cervical or elbow lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
muscular activity | 6 and 12 weeks post surgery
  Activity of upper trapezius, anterior, middle and posterior parts of deltoid ans of infraspinatus.
  The mean amplitude of electromyographic (EMG) signal, expressed as a percentage of reference voluntary contraction (RVC) is used

SECONDARY OUTCOMES:
active range of motion | 6 and 12 weeks post surgery
  shoulder flexion measured in degrees
strength | 6 and 12 weeks post surgery
  isometric strength at 90° of shoulder flexion, measured in kg
pain | 6 and 12 weeks post surgery
  shoulder pain intensity measured with a 100-mm visual analog scale (0: no pain; 100: worst imaginable pain). Shoulder pain intensity was assessed at end-point of ROM and after isometric force assessment. This measure is known for its excellent reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Léger, PhD, Study Chair — Clinique romande de réadaptation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kase K, Wallis J, Kase T: Clinical Therapeutic Applications of the Kinesio Taping Method. Tokyo, Japan: Keni-Kai information; 2003.
- [Derived] Reynard F, Vuistiner P, Leger B, Konzelmann M. Immediate and short-term effects of kinesiotaping on muscular activity, mobility, strength and pain after rotator cuff surgery: a crossover clinical trial. BMC Musculoskelet Disord. 2018 Aug 22;19(1):305. doi: 10.1186/s12891-018-2169-5. PMID 30134883